CLINICAL TRIAL: NCT07233512
Title: EFFECT OF SURGICAL AND NON-SURGICAL PERIODONTAL TREATMENT ON ALZHEIMER DISEASE-ASSOCIATED OUTCOMES: A Randomized Clinical Trial
Brief Title: EFFECT OF PERIODONTAL TREATMENT ON ALZHEIMER DISEASE-ASSOCIATED OUTCOMES
Acronym: PETAL
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Liege (Other)
Collaborators: Eklund foundation Malmö (Unknown)
Responsible Party: Principal Investigator, Altaep Yaman, Periodontist - Oral surgeon, Centre Hospitalier Universitaire de Liege
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: B7072021000057
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Alzheimers Disease; Periodontitis
Keywords: Alzheimer's disease; periodontitis; neuroinflammation; randomized controlled trial; cognitive function
MeSH Terms: conditions — Alzheimer Disease; Periodontitis; Neuroinflammatory Diseases

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TEST GROUP (Experimental): Test group: 35 patients diagnosed with both mild to moderate stage of AD and periodontal disease.This group will receive immediatly complete periodontal treatment: an initial periodontal therapy (step 1 and 2) along with any needed dental extractions, and with an intensive supportive periodontal care follow-up (every 3 months). At 12 months from baseline, patients will receive an additional periodontal surgical therapy (step 3 of periodontal therapy). and/or an intensive supportive periodontal care (SPC) follow-up every 3 months (step 4)
  Interventions: Procedure: INITIAL PERIODONTAL THERAPY
- CONTROL GROUP (Active Comparator): o Control group: 35 patients diagnosed with both mild to moderate stage of AD and periodontal disease. This group will receive a delayed periodontal therapy (step 1, 2, and 3 ) 6 months after the test group along with a regular supportive periodontal care follow-up (every 6 months). At 12 months from baseline, patients will receive an additional periodontal surgical therapy (step 3 of periodontal therapy) and/or an intensive supportive periodontal care (SPC) follow-up every 3 months (step 4)
  Interventions: Procedure: INITIAL PERIODONTAL THERAPY
- COMMON GROUP (Experimental): At the 12-month mark, all participants-regardless of initial group allocation-will be merged into a single cohort. At this stage, additional periodontal surgical therapy (Step 3) will be administered, followed by intensified supportive periodontal care (Step 4), consisting of maintenance visits every 3 months for the remainder of the study period.
  Interventions: Procedure: INITIAL PERIODONTAL THERAPY

INTERVENTIONS:
Procedure: INITIAL PERIODONTAL THERAPY — The intervention will be an initial periodontal therapy (step 1 and 2). Instrumentation will be performed by two calibrated periodontists (Y.A. & L.S) using an ultrasonic piezoelectric device with specific micro-inserts (Newtron P5 XS Bled, Acteon, Satelec, France). Local subgingival disinfection will be performed using hydrogen peroxide and povidone iodine 1%. The patients will be trained to maintain good personal oral hygiene, including interdental hygiene (floss, brushes) and water for chemical plaque control containing 0.2% chlorhexidine, 3 - 4 weeks twice a day. This initial periodontal therapy will be carried out at different time points depending on the group (test group and control group).The initial periodontal therapy also include extractions of hopeless teeth. A clinical reevaluation will be conducted three months after completion of the initial periodontal therapy in the test group, and twelve months after baseline in the control group.
  Other Names: HOPELESS TOOTH EXTRACTION; ADDITIONAL PERIODONTAL SURGICAL THERAPY

SUMMARY:
Periodontitis is the most prevalent chronic infectious inflammatory disease in adults, leading to the destruction of tooth-supporting tissues. Beyond its local impact, periodontitis contributes to systemic inflammation through the release of periodontal pathogens and their byproducts into the bloodstream. Given that chronic intracerebral inflammation is a known driver of Alzheimer's disease (AD) progression, a biological link between the two conditions has been hypothesized. This study aims to evaluate whether periodontal treatment can influence AD progression by reducing systemic inflammation. We have designed a randomized controlled clinical trial including 70 patients diagnosed with both AD and stage 3 or 4 periodontitis, randomly allocated to receive either immediate (test group) or delayed (control group) periodontal therapy. All participants will undergo comprehensive periodontal treatment and be followed over a 24-month period. Cognitive assessments, periodontal evaluations, blood and saliva biomarker analyses, and neuroimaging will be conducted at multiple time points to assess the potential impact of periodontal therapy on AD progression. This trial represents the first clinical investigation into the effect of periodontal treatment on the course of Alzheimer's disease.

DETAILED DESCRIPTION:
Impact of Periodontal Treatment on Alzheimer's Disease Progression (PETAL Study)

**Study Overview** This randomized controlled clinical trial aims to investigate the impact of comprehensive periodontal treatment on cognitive, functional, biomarker, and neuroinflammatory outcomes in patients with mild to moderate Alzheimer's disease (AD) presenting advanced periodontitis. The study evaluates whether the reduction of oral and systemic inflammation through periodontal therapy can influence the progression of Alzheimer's disease. The trial will be conducted at the University Hospital of Liège, Belgium, under the collaboration between the Departments of Neurology and Periodontology. The project is titled PETAL (Periodontal Treatment in Alzheimer's Disease) and will recruit seventy participants over a 24-month follow-up period.

**Background and Rationale** Alzheimer's disease is a chronic neurodegenerative condition characterized by progressive decline in cognitive and memory functions, ultimately leading to functional impairment and loss of independence. The disease is associated with the accumulation of amyloid-beta plaques and neurofibrillary tangles, synaptic dysfunction, and neuroinflammation. Periodontitis, a chronic inflammatory disease affecting the supporting structures of the teeth, is a highly prevalent condition that induces local and systemic inflammation through the dissemination of periodontal pathogens and their by-products into the bloodstream. Increasing evidence supports a bidirectional relationship between chronic periodontitis and systemic conditions, including diabetes, cardiovascular disease, and neurodegenerative disorders such as Alzheimer's disease. Inflammatory mediators derived from periodontal infection may contribute to neuroinflammatory processes that exacerbate neuronal injury and cognitive decline.

The proposed biological mechanism linking periodontitis and Alzheimer's disease involves the entry of periodontal bacteria and their toxins into systemic circulation, triggering immune responses that elevate levels of inflammatory cytokines such as IL-1β, IL-6, TNF-α, and CRP. These mediators can cross the blood-brain barrier, contributing to microglial activation and neuroinflammation. Pathogens like *Porphyromonas gingivalis* and their virulence factors (gingipains) have been detected in brain tissue, supporting a mechanistic link. Preclinical studies have shown that periodontal infection may increase amyloid-beta production, activate the complement cascade, and promote neurodegeneration. Therefore, periodontal therapy aimed at reducing bacterial load and systemic inflammation could potentially attenuate Alzheimer's-related pathology.

**Objectives** The primary objective is to determine whether initial non-surgical periodontal therapy combined with intensive supportive periodontal care improves cognitive performance and neuroinflammatory biomarkers in patients with Alzheimer's disease and advanced periodontitis. The secondary objective is to evaluate whether additional periodontal surgical therapy followed by intensive supportive periodontal care enhances cognitive and biological outcomes over 24 months.

**Study Design** This is a single-center, randomized, controlled, parallel-group clinical trial including seventy patients diagnosed with mild-to-moderate Alzheimer's disease and stage 3 or 4 periodontitis. Participants will be randomly assigned to either an immediate treatment group (test) or a delayed treatment group (control). The control group will begin periodontal therapy six months later than the test group. All patients will undergo comprehensive periodontal and cognitive assessments, biomarker analyses, and neuroimaging at multiple time points during the 24-month study period.

At baseline, both groups will undergo clinical, cognitive, and biological evaluations. The test group will receive immediate periodontal therapy consisting of steps 1 and 2 (behavioral modification, supra- and sub-gingival instrumentation, and extraction of hopeless teeth) followed by intensive supportive periodontal care every three months. The control group will receive the same treatment six months later, with regular supportive care every twelve months during the first year. After twelve months, both groups will receive additional periodontal surgical therapy (step 3) and continue with intensive supportive periodontal maintenance (step 4) every three months until the end of the study.

**Sample Size and Statistical Considerations** Sample size calculations were based on detecting a 0.9 z-score difference in the Preclinical Alzheimer Cognitive Composite (PACC), assuming a standard deviation of 1.0, a 90% power, and a 2.5% significance level to account for multiple hypotheses testing. Accounting for a 10% dropout rate, a total of 70 participants (35 per group) will be enrolled. Data will be analyzed using mixed-effects models for repeated measures, comparing changes in cognitive, functional, periodontal, and biomarker outcomes between groups across time points.

**Interventions**

Periodontal treatment will follow a standardized four-step approach:

Step 1: Behavioral modification, supragingival plaque control, and risk factor management.

Step 2: Non-surgical supra- and subgingival instrumentation using ultrasonic piezoelectric devices, with local disinfection using hydrogen peroxide and povidone iodine.

Step 3: Periodontal surgical therapy (if indicated) to treat residual pockets and achieve optimal tissue health.

Step 4: Supportive periodontal care (SPC) every three months, including professional cleaning and reinforcement of oral hygiene instructions.

All treatments will be performed by calibrated periodontists using standardized protocols. Patients will receive individualized oral hygiene instructions and prescribed electric toothbrushes and interdental brushes. The goal is to reduce periodontal pocket depth, bleeding on probing, and plaque accumulation, thereby minimizing systemic inflammatory burden.

**Outcome Measures**

Primary Outcome:

- Cognitive status assessed by the Preclinical Alzheimer Cognitive Composite (PACC), integrating memory, executive, and global cognitive function scores.

Secondary Outcomes:

* Functional ability measured by the Disability Assessment for Dementia (DAD-6).
* Burden of disease in daily activities for patient and caregiver.
* Periodontal health indices, including probing depth, clinical attachment level, bleeding on probing, furcation involvement, and plaque score.
* Biomarkers: Amyloid-beta (Aβ40, Aβ42), phosphorylated tau protein, and inflammatory cytokines in blood and saliva.
* Neuroimaging outcomes: brain gray matter volume and hippocampal subfield mapping using MRI.

**Eligibility Criteria**

Inclusion criteria:

* Clinical diagnosis of probable Alzheimer's disease (NIA-AA criteria).
* Mild to moderate cognitive impairment (MMSE >15).
* Stage 3 or 4 periodontitis with at least 10 residual teeth.
* No contraindications to MRI.
* Signed informed consent from patient or legal representative.

Exclusion criteria:

* Participation in another clinical trial within the past 30 days.
* Antibiotic use in the past three months.
* Immunosuppressive therapy or chemotherapy.
* Contraindications to MRI or inability to undergo imaging.

**Data Collection and Analysis** Cognitive and functional data will be obtained through standardized neuropsychological assessments. The PACC will evaluate global cognitive performance using z-scores derived from memory recall, digit symbol substitution, category fluency, and MMSE results. Functional independence will be measured with DAD-6, and caregiver burden will be scored from 0 to 3. Periodontal data will include probing depth, attachment loss, plaque index, bleeding on probing, and furcation involvement. Blood and saliva samples will be collected for biomarker quantification and stored at -80°C. Neuroimaging will assess brain atrophy and gray matter volume using 3T MRI, analyzed with the SPM12 Longitudinal Toolbox.

Biological analyses will include ELISA quantification of amyloid-beta peptides and phosphorylated tau, and multiplex immunoassays for inflammatory cytokines (IL-1β, IL-6, IL-10, TNF-α, CRP). Microbiological analysis will involve 16S rDNA sequencing to assess subgingival microbiome composition, processed through DADA2 and LEfSe pipelines to identify taxa associated with systemic inflammation and cognitive decline.

**Study Significance** This study is among the first randomized controlled clinical trials to directly evaluate the causal impact of periodontal therapy on Alzheimer's disease progression. It integrates advanced cognitive testing, biomarker profiling, and neuroimaging to explore how oral inflammation influences neurodegeneration. By identifying whether controlling periodontal disease can reduce systemic inflammation and slow cognitive decline, this research may open new preventive and therapeutic pathways linking oral and brain health.

**Ethical and Regulatory Considerations** The study has been approved by the Human Research Ethics Committee of the University Hospital of Liège. Written informed consent will be obtained from all participants or their legal representatives. All data will be anonymized and handled in accordance with the General Data Protection Regulation (GDPR). The study will be registered on ClinicalTrials.gov prior to participant enrollment.

**Conclusion** The PETAL study will provide critical insights into the relationship between chronic periodontal inflammation and Alzheimer's disease pathology. If periodontal treatment demonstrates a beneficial effect on cognitive or biological outcomes, it would support a novel, non-pharmacological, and accessible intervention to improve quality of life and slow the progression of neurodegenerative diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Have to suffer from AD
2. Must agree to have brain imaging (without contra-indication for MRI)
3. Possess a minimum of 10 residual teeth
4. Have an MMSE score greater than 15
5. Exhibit a DPSI score of ≥ 3+ indicating advanced periodontal disease

Exclusion Criteria:

1. Participation in another clinical trial (30 days)
2. Contra-indication for MRI
3. Use of antibiotics in the past 3 months
4. Immunosuppressive drugs or chemotherapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2023-11-17 (Actual); Primary Completion 2029-09-10 (Estimated); Study Completion 2029-09-10 (Estimated)

PRIMARY OUTCOMES:
Cognitive status using pre-clinical Alzheimer cognitive composite (PACC) | From enrollment to the end of the study at 24 months for the test group. And from 6 months until the end of the study at 24 months
  The Preclinical Alzheimer Cognitive Composite (PACC) is a sensitive neuropsychological tool designed to detect subtle cognitive decline in the early stages of Alzheimer's disease (AD). It combines several tests assessing memory, executive function, and global cognition, including the Free and Cued Selective Reminding Test (FCSRT), Logical Memory delayed recall, Digit Symbol Substitution Test, and Mini-Mental State Examination. Each test score is standardized into z-scores and averaged to produce a composite reflecting global cognition. The PACC is validated as a primary outcome measure in AD prevention trials, showing strong correlations with amyloid and tau biomarkers, and enabling early detection of cognitive decline before dementia onset.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Liège, Université de Liège Domaine du Sart Tilman, Liège, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Stein PS, Desrosiers M, Donegan SJ, Yepes JF, Kryscio RJ. Tooth loss, dementia and neuropathology in the Nun study. J Am Dent Assoc. 2007 Oct;138(10):1314-22; quiz 1381-2. doi: 10.14219/jada.archive.2007.0046. PMID 17908844
- [Result] Querfurth HW, LaFerla FM. Alzheimer's disease. N Engl J Med. 2010 Jan 28;362(4):329-44. doi: 10.1056/NEJMra0909142. No abstract available. PMID 20107219
- [Result] Perry VH, Newman TA, Cunningham C. The impact of systemic infection on the progression of neurodegenerative disease. Nat Rev Neurosci. 2003 Feb;4(2):103-12. doi: 10.1038/nrn1032. No abstract available. PMID 12563281
- [Result] Farhad SZ, Amini S, Khalilian A, Barekatain M, Mafi M, Barekatain M, Rafei E. The effect of chronic periodontitis on serum levels of tumor necrosis factor-alpha in Alzheimer disease. Dent Res J (Isfahan). 2014 Sep;11(5):549-52. PMID 25426144
- [Result] Kamer AR, Craig RG, Pirraglia E, Dasanayake AP, Norman RG, Boylan RJ, Nehorayoff A, Glodzik L, Brys M, de Leon MJ. TNF-alpha and antibodies to periodontal bacteria discriminate between Alzheimer's disease patients and normal subjects. J Neuroimmunol. 2009 Nov 30;216(1-2):92-7. doi: 10.1016/j.jneuroim.2009.08.013. Epub 2009 Sep 19. PMID 19767111
- [Result] Costa MJF, de Araujo IDT, da Rocha Alves L, da Silva RL, Dos Santos Calderon P, Borges BCD, de Aquino Martins ARL, de Vasconcelos Gurgel BC, Lins RDAU. Relationship of Porphyromonas gingivalis and Alzheimer's disease: a systematic review of pre-clinical studies. Clin Oral Investig. 2021 Mar;25(3):797-806. doi: 10.1007/s00784-020-03764-w. Epub 2021 Jan 20. PMID 33469718
- [Result] Carter CJ, France J, Crean S, Singhrao SK. The Porphyromonas gingivalis/Host Interactome Shows Enrichment in GWASdb Genes Related to Alzheimer's Disease, Diabetes and Cardiovascular Diseases. Front Aging Neurosci. 2017 Dec 12;9:408. doi: 10.3389/fnagi.2017.00408. eCollection 2017. PMID 29311898
- [Result] Dioguardi M, Caloro GA, Troiano G, Giannatempo G, Laino L, Petruzzi M, Lo Muzio L. Oral manifestations in chronic uremia patients. Ren Fail. 2016;38(1):1-6. doi: 10.3109/0886022X.2015.1103639. Epub 2015 Oct 29. PMID 26513593
- [Result] Heimdahl A, Hall G, Hedberg M, Sandberg H, Soder PO, Tuner K, Nord CE. Detection and quantitation by lysis-filtration of bacteremia after different oral surgical procedures. J Clin Microbiol. 1990 Oct;28(10):2205-9. doi: 10.1128/jcm.28.10.2205-2209.1990. PMID 2229342
- [Result] Tatakis DN, Kumar PS. Etiology and pathogenesis of periodontal diseases. Dent Clin North Am. 2005 Jul;49(3):491-516, v. doi: 10.1016/j.cden.2005.03.001. PMID 15978238
- [Result] Haffajee AD, Socransky SS. Introduction to microbial aspects of periodontal biofilm communities, development and treatment. Periodontol 2000. 2006;42:7-12. doi: 10.1111/j.1600-0757.2006.00190.x. No abstract available. PMID 16930302
- [Result] Kumar A, Singh A, Ekavali. A review on Alzheimer's disease pathophysiology and its management: an update. Pharmacol Rep. 2015 Apr;67(2):195-203. doi: 10.1016/j.pharep.2014.09.004. Epub 2014 Sep 22. PMID 25712639
- [Result] Venneti S, Wang G, Nguyen J, Wiley CA. The positron emission tomography ligand DAA1106 binds with high affinity to activated microglia in human neurological disorders. J Neuropathol Exp Neurol. 2008 Oct;67(10):1001-10. doi: 10.1097/NEN.0b013e318188b204. PMID 18800007
- [Result] Schwab C, McGeer PL. Inflammatory aspects of Alzheimer disease and other neurodegenerative disorders. J Alzheimers Dis. 2008 May;13(4):359-69. doi: 10.3233/jad-2008-13402. PMID 18487845
- [Result] Gaur S, Agnihotri R. Alzheimer's disease and chronic periodontitis: is there an association? Geriatr Gerontol Int. 2015 Apr;15(4):391-404. doi: 10.1111/ggi.12425. Epub 2014 Dec 16. PMID 25511390